CLINICAL TRIAL: NCT04513977
Title: Geriatric Oncology SuPportive Clinic for ELderly
Acronym: GOSPEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Goh Wen Yang (Other)
Collaborators: The Palliative Care Centre for Excellence in Research and Education (PalC) (Unknown); Lee Kong Chian School of Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Goh Wen Yang, Consultant, Tan Tock Seng Hospital
Organization: Tan Tock Seng Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DSRB: 2019/00639
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Frailty
Keywords: Geriatric Oncology; Frailty; Comprehensive Geriatric Assessment; Quality of life
MeSH Terms: conditions — Neoplasms; Frailty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): For older adults with cancer with G8 score 14 or less. Randomized to usual oncology care.
- Geriatric Oncology Supportive Clinic (Experimental): For older adults with cancer with G8 score 14 or less. Randomized to attend Geriatric Oncology Supportive Clinic
  Interventions: Other: Geriatric Oncology Supportive Clinic

INTERVENTIONS:
Other: Geriatric Oncology Supportive Clinic — Patients will undergo Comprehensive Geriatric Assessment with subsequent tailored intervention based on deficits identified. Comprehensive palliative assessment for any symptom burden and symptommatic treatment will be done as well.
  Arms: Geriatric Oncology Supportive Clinic

SUMMARY:
This is a randomized controlled trial comparing the impact of Geriatric-Oncology-Supportive Clinic (GOSC) on quality of life in older adult with newly diagnosed cancer undergoing cancer related treatment.

DETAILED DESCRIPTION:
(i) Recognition of unique need of older adults cancer patients Cancer is a disease largely affecting the older adults, with incidence of malignancies after age of 65 years 11 folds higher than younger adults. Despite this, our understanding of cancer treatment effects in older adults is poor because they are largely unrepresented in such trials. Efforts to extrapolate cancer treatment effects from younger adults to the older adults have been difficult because of their heterogeneous health status, which lead to a recognition of the need for Comprehensive Geriatric Assessment (CGA) to detect vulnerability and formulate individualized care plan. This awareness has been echoed in multiple international guidelines including the American Society of Clinical Oncology (ASCO), European Organization for Research and Treatment of Cancer (EORTC), European Society of Medical Oncology (ESMO), National Comprehensive Cancer Network (NCCN) and has led to the founding of International Society of Geriatric Oncology (SIOG) in 2000.

(ii) Geriatric-Oncology In Geriatric Medicine, CGA is the cornerstone in caring for the older adults and is defined as "multidisciplinary diagnostic and treatment process that identifies medical, psychosocial, and functional capabilities of older adults to develop a coordinated plan to maximize overall health with aging". The diagnostic outcomes and treatment targets of CGA are traditionally represented as "geriatric giants" including instability, incontinence, immobility and intellectual impairment, with recent inclusion of "modern geriatric giants" represented by frailty and sarcopenia. CGA has been shown to improve function, health status, quality of life and healthcare utilization outcomes in diverse clinical settings. It is important to understand that the key to improve patient outcomes based on CGA relies not only on the assessment butalso the intervention that follows. The CGA by a geriatrician, however, is labor-intensive, time consuming and limited by the number of geriatricians available. Hence, in a busy oncology clinic, there are 3 recommended approaches for assessment of older adults. Firstly, in a form of risk assessment tool, such as Cancer and Aging Research Group (CARG) or Chemotherapy Risk Assessment Scale for High-Age Patients (CRASH), that predicts likelihood of toxicity from chemotherapy. Secondly, a screening test, such as Geriatric-8 (G8) with an aggregate that serves to identify vulnerable older adults who may benefit from a subsequent CGA. Thirdly, a geriatric assessment (GA) which takes into account the different domains of CGA to identify vulnerable older adults who may benefit from a subsequent CGA. The above 3 pathways also form the current models of care for geriatric-oncology. G8 has been recommended by ASCO and EORTC as a screening test of choice (<=14 as vulnerable and >14 as fit) with good sensitivity, specificity, positive predictive value and negative predictive value for vulnerability against CGA assessment outcomes as the gold standard. G8 has been extensively studied in older adults with cancer undergoing radio(chemo)therapy.

(iii) Special consideration to older adults with early and locally advanced cancer Current published trials and ongoing trials focused on older adults who are undergoing oncological treatment regardless on cancer stage. However, generally, early and locally advanced cancer patients and advanced cancer groups should not be regarded to be homogenous. Firstly, the intention for treatment may be vastly different with most of the advanced cancer group being treated with palliative intent. Henceforth, the treatment intensity, frequency and likelihood for further treatment escalation is higher in early and locally advanced cancer. Secondly, the prognosis between the 2 groups, in view of disease burden and treatment intent, will be vastly different. Thirdly, recently studies of early palliative care has shown significant improvement in quality of life and mood in patients with advanced cancer, but there had been no studies looking at early and locally advanced cancer group. Henceforth, older adults with early and locally advanced cancer is a unique group facing higher potential of complication from treatment with worsened quality of life for a prolonged period of life without any useful service option.

(iv) Special consideration to early palliative care in older adults with newly diagnosed cancer In older adults, frequently their focus is for maintenance of quality of life and less so for prolonging life. In Geriatric-Oncology, this aim is fulfilled by (1) detecting vulnerability (2) intervention to maintain fitness and quality of life (3) providing advice to oncologist for optimized management. However, we propose for a 4th dimension of care for older adults with cancer which entails symptom control from principles of palliative care. It is crucial to know that poorly controlled symptoms is associated with poorer quality of life. This is even more important for older adults who are not undergoing treatment. Henceforth, to look into maintenance of quality of life, there had been recent calls for integration of palliative care with geriatric oncology.

(v) Identified evidence gap Despite multiple studies looking at the efficacy of Geriatric-Oncology, there had been a paucity in research on its impact on quality of life. This is especially so specifically for older adults with early and locally advanced cancer who may suffer for a prolonged time with poor quality of life. Research is also lacking on the effect of palliative care in early and locally advanced cancer. Henceforth the impetus to seek for the benefit of a new service that integrates principles of Geriatric-Oncology with palliative care.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and above
* Newly diagnosed early or locally advanced cancer
* Planned for treatment

  * high dose radiotherapy (both curative and palliative) and / or
  * curative chemotherapy

Exclusion Criteria:

* Seen in Geriatric or Palliative Medicine Clinic in prior 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
HRQOL questionnaire (EORTC QLQ-ELD14) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wen Yang Goh, Principal Investigator — TTSH
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goh WY, Tan HM, Teo HL, Vong EKY, Ho FCH, Lim MY, Hum AYM. Clinical Frailty Scale versus Geriatric-8 in predicting quality of life among older adults receiving curative cancer treatment. Support Care Cancer. 2025 Jun 6;33(7):550. doi: 10.1007/s00520-025-09616-1. PMID 40478269
- [Derived] Goh WY, Neo HY, Teo HL, Koh MYH, Griva K, Lim MY, Ho FCH, Hum AYM. Protocol for a randomised controlled trial on impact of comprehensive geriatric and supportive assessment versus standard care in older adults with cancer undergoing curative treatment: The Geriatric Oncology SuPportive clinic for ELderly (GOSPEL) study. J Geriatr Oncol. 2023 Jan;14(1):101342. doi: 10.1016/j.jgo.2022.07.002. Epub 2022 Jul 15. PMID 35843845